CLINICAL TRIAL: NCT03445221
Title: Implication of Preoperative Immunonutrition Upon Cardiac Patients Undergoing Mitral Valve Replacement Surgery
Brief Title: Preoperative Immunonutrition and Cardiac Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed F. Mostafa, Associate Professor of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Immunonutrition
Record Dates: First submitted 2018-02-16; First posted 2018-02-26 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Function
Keywords: Immunonutrition; Cardiac Patient; Mitral Valve Replacement
MeSH Terms: interventions — Immunonutrition Diet

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Patients will receive preoperative immunonutrition in the form of glutamine) Dipeptiven-Fresenius Kabi) given by intravenous infusion 0.4g/kg/day for 3 days before surgery.
  Interventions: Dietary Supplement: IV Immunonutrition
- Group II (Active Comparator): Patients will continue preoperative oral conventional diet.
  Interventions: Dietary Supplement: Conventional Diet

INTERVENTIONS:
Dietary Supplement: IV Immunonutrition — patients will receive preoperative immunonutrition in the form of glutamine) Dipeptiven-Fresenius Kabi) given by intravenous infusion 0.4g/kg/day for 3 days before surgery.
  Arms: Group I
Dietary Supplement: Conventional Diet — patients will continue preoperative oral conventional diet.
  Arms: Group II

SUMMARY:
With the progress of cardiac surgery, the indication of cardiac valve replacement has been extended to include severely ill patients, even those with cardiac cachexia caused by long-standing mitral valve disease. Since patients with advanced cardiac functional disability are prone to fall into a low cardiac output state after valve replacement, Those severely ill, cachectic patients may be susceptible to postoperative acute renal failure. Preoperative malnutrition because of poor oral intake significantly increases the risk of adverse events after surgery and leads to increased length of stay.

Major operation itself possibly cause the dysfunction of the host homeostasis, defense mechanisms and inflammatory response, which would increase the rate of postoperative complications and prolong hospital stay. Recently, many researchers argued that immunonutritional formulas supplemented with biologically active nutrients were more effective than standard nutrition intervention in improving inflammation, promoting the wound healing and shortening the length of hospital stay (LOS) after operation.

DETAILED DESCRIPTION:
Eligibility and type of the study: This randomized clinical trial will be conducted at Assiut University Hospital from March 2018 until March 2019 after approval from the Institutional Ethics Committee and after obtaining written informed consents from all cardiac patients undergoing mitral valve replacement surgery.

Randomization and sample size :

Sample size calculation Sample size calculation was carried out using G*Power 3 software. A calculated sample of 88 patients (44 cases and 44 controls) will be needed to detect an effect size of 0.3 reduction in pro-BNP Level, with an error probability of 0.05 and 90% power on a two-tailed test.

Patients:

Patients will be assigned into two equal groups of 44 patients each:

Group 1: patients will take preoperative immunonutrition in the form of intravenous glutamine (Dipeptiven-Fersenius Kabi) 0.4 g/kg/day (once daily) for 5 days before surgery in addition to a conventional diet.

Group 2: patients will continue conventional diet. Conventional median sternotomy will be performed in all patients. Arterial line will be inserted. Anesthesia will be induced with midazolam 0.05mg\kg, propofol 1-1.5mg\kg and fentanyl 2μg\kg. Anesthesia will be maintained with isoflurane, fentanyl infusion1-2μ\kg\hr and Cis-atracurium infusion 2μ\kg\min before cardiopulmonary bypass (CBP) and with propofol and fentanyl on CBP, according the anaesthetist criteria. Anticoagulation will be achieved with heparin 3-4 mg\kg to maintain an activated clotting time over 450s .Reversal of heparin will be with protamine. Cardiopulmonary bypass will be achieved with a roller pump and a membrane oxygenator. After the aortic clamp will be applied, asolution of 1000-1500 cc of hematic cardioplegia will be administrated. Then 400-500 cc of solution will be administrated every 30min until the end of the procedure. Mean arterial pressure should be above 60 mmHg for the duration of CBP.

Data collection:

Cardiac function:

* Preoperative and postoperative echocardiography.
* Inotropic score every 2hours in first 6 hours then every 6 hours for the rest of 48 hours postoperatively.
* Serum proBNP (Brain natruritic peptide) preoperatively and post operative first and forth days.

Kidney function:

* Urine output in the postoperative first and second days.
* Serum urea and creatinine in postoperative first and second days.
* Serum NGAL (Neutrophil gelatinase-associated lipocalin) preoperatively and postoperative first and forth days.

Hemodynamics:

- MAP, HR every 2hours in first 6 hours then every 6 hours for the rest of 48 hours postoperatively.

Hours of mechanical ventilation. Hospital and ICU stay. Any postoperative complications will be recorded and treated.

Sampling:

Venous blood sample will be obtained by direct venipuncture and collected into serum separator tubes. Samples will be centrifuged within 20 minutes from withdrawal and stored for amixture of 12 hours at 2-8 ゜C before the separation of serum. Serum will be stored frozen at -40 ゜C. Pro-BNP serum concentrations will be determined using an automated method.

Statistical analysis :

Data will be performed using a standard SPSS software package version 21 (SPSS Inc., Chicago, Illinois, USA).Descriptive values will be expressed as mean ± SD, number or percentages. The Student t-test will be used for comparison between means of variables and normally distributed data. P will be considered significant if (p≤ 0.05).

Ethical Consideration:

* The randomized clinical trial will be approved by local ethics committee of faculty of medicine, Assiut University, Egypt after obtaining written informed consent from patients.
* There is no risk affecting the patients participating in this study.
* Every patient can leave the study and will receive the same care.
* Any data taken from all patient will be made confidential and available only to persons conducting the study.
* Any patient can stop participation in the study at any time without any loss of service.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Age: 18-60 years.
* Valvular heart disease .
* ASA II,III
* Non-diabetic.
* Elective surgery.

Exclusion Criteria:

* Pre-existing renal disease(creatinine3.5mg/dl or dialysis)
* Diabetic.
* Off pump surgery.
* Long CBP time >120 min .
* Previous cardiac surgery.
* Hepatic failure or established cirrhosis.
* Emergency surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Cardiac Fuction | 4 days
  Serum proBNP (Brain natruritic peptide)

SECONDARY OUTCOMES:
Inotropic score | 4 days
  Dopamine dose (mcg/kg/min) + Dobutamine dose (mcg/kg/min) + 100 x Epinephrine dose (mcg/kg/min) min 20 and max 60 The lower the inotropic score the better cardiac function and lower morbidity
Kidney Function | 4 days
  Serum NGAL (Neutrophil gelatinase-associated lipocalin)
urine output | 2 days
  urine volume per day
Hemodynamics | 2 days
  mean arterial blood pressure
Postoperative Hospital Data | 4 days
  Hospital and ICU stay
Postoperative complications | 4 days
  any postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Khaled M Morsy, MD, Study Director — Assistant prof of anesthesia and intensive care
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided